CLINICAL TRIAL: NCT03994354
Title: Taipei Medical University Shuang-Ho Hospital
Brief Title: The Wound Infection After Stomy Closure Between Different Methods of Drainage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, Chief of colorectal surgery, Taipei Medical University Shuang Ho Hospital
Other Study IDs: N201905015
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Wound Infection
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1,2: 1. J-P drain group
  2. Penrose drain group
  Interventions: Procedure: J-P drainage and cutaneous penrose drainage insertion

INTERVENTIONS:
Procedure: J-P drainage and cutaneous penrose drainage insertion — Lots of the stoma wound closure technique have been developed, including subcutaneous antibiotic material implantation, wound irrigation with iodine, closure wound with a drain tube, secondary closure, delayed primary closure and pursestring closure. But there still is in debate about best skin closure test. In Division of Colorectal Surgery Shuang Ho Hospital, two current stoma wound closure methods were subcutaneous Jackson-Pratt drainage and cutaneous penrose drainage insertion.

SUMMARY:
This proposal will investigate the wound condition between different drainage methods of the stoma closure wound. Anastomotic leakage is a major complication after colorectal surgery. The protective stoma will decrease the anastomosis leakage rate and severity1. Stoma closure is often performed after the condition of the previous protecting site improved. Wound infection is not a rare complication after stoma closure, with a reported infectious rate from 3% to 43%. Wound infection will result in wound dehiscence, incisional herniation, ileus and the length of hospital stay. Lots of the stoma wound closure technique have been developed, including subcutaneous antibiotic material implantation, wound irrigation with iodine, closure wound with a drain tube, secondary closure, delayed primary closure and pursestring closure. But there still is in a debate about the best skin closure test. In Division of Colorectal Surgery Shuang Ho Hospital, two current stoma wound closure methods were subcutaneous Jackson-Pratt drainage and cutaneous Penrose drainage insertion.

In the project, clinical outcomes of these two drainage methods will be compared. The subcutaneous. Jackson-Pratt drainage is used to create negative pressure in subcutaneous closure wound. The negative pressure will extract actively the tissue debris and fluid, avoiding the seroma and pus accumulation. The cutaneous Penrose drainage is used to create delayed skin healing, and the tissue debris and fluid will drainage passive by capillary phenomenon. Two groups will be distributed randomly. The demographic characters like age, gender, BMI, nutritional status, under chemotherapy, diabetes and past medication history will be reviewed. Perioperative clinical data like the method of the anastomosis, operation time, postoperative hospital day, surgical site infection, prolonged ileus, anastomosis leakage, and incisional hernia will be collected.

From this study, these two stoma wound closure methods will be evaluated and analyze the risk factors of complication for the stoma wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered from colon or ileum stoma. After the doctor's evaluation, the distal bowel tract was normal.

Exclusion Criteria:

* Pregnancy, child, psychiatric disorder, behavior disorder, and prisoner. And those patients can't follow the protocol

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who had suffered from colostomy or ileostomy in previous operation will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2019-07-06 (Actual); Primary Completion 2022-07-07 (Estimated); Study Completion 2022-07-07 (Estimated)

PRIMARY OUTCOMES:
Wound infection | Wound infection in post-operation 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan